CLINICAL TRIAL: NCT01063010
Title: Pilot Study of Bevacizumab (Avastin) in Patients With Septic Shock
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: The Cooper Health System (Other); Carolinas Medical Center (Other)
Responsible Party: Principal Investigator, Nathan Shapiro, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009000036
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Septic Shock
Keywords: sepsis; septic shock; Bevacizumab; Avastin
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo IV for 90 minutes (+ 15 minutes)
  Interventions: Drug: Placebo
- Bevicizumab (Experimental): IV infusion over 90 minutes
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Administered intravenously 10 mg/kg over 90 minutes (+ 15 minutes)
  Other Names: Avastin
  Arms: Bevicizumab
Drug: Placebo — Placebo administered intravenously for 90 minutes (+ 15 minutes)
  Arms: Placebo

SUMMARY:
The purpose of this study is to perform a pilot study to assess the potential use of Bevacizumab (a vascular endothelial growth factor (VEGF) inhibitor) in sepsis.

DETAILED DESCRIPTION:
Sepsis is responsible for significant morbidity, mortality, and costs to patients in our healthcare system. The hospital case mortality rate for severe sepsis (sepsis with acute organ system dysfunction) is between 30-50%,7-12 with an incidence of approximately 751,000 cases and 215,000 deaths nationally per year. The overall cost of care is estimated at $16.7 billion annually in the US.Despite significant advances in medical science, the overall mortality rate for severe sepsis has not improved substantially over time.

VEGF signaling and sepsis. VEGF contributes to inflammation and coagulation - the key elements in sepsis pathophysiology. For example, under in vitro conditions, VEGF induces the expression of cell adhesion molecules (E-selectin, ICAM-1, and VCAM-1) in endothelial cells and promotes adhesion of leukocytes. Moreover, VEGF signaling upregulates tissue factor mRNA, protein and procoagulant activity. Several studies have shown increased circulating levels of VEGF in patients with sepsis. In one study, maximum VEGF levels were increased in survivors versus non-survivors in sepsis. In another study of patients with meningococcal meningitis, elevated VEGF levels were associated with shock and upregulation of IL-1beta, IL-10, IL-12, complement activation and increased permeability.We have additional human data on 83 patients demonstrating an association of VEGF with SOFA score, IL-1, and IL-6. Consistent with its critical role in inflammation, VEGF inhibition using a VEGF trap resulted in attenuation of plasma interleukin IL-6 and IL-10 levels in a mouse cecal ligation puncture (CLP) model.

VEGF signaling is an important determinant of sepsis morbidity and mortality in animal models. We have recently shown that sepsis is associated with a time-dependent increase in circulating levels of VEGF in animal and human models of sepsis.2 The overexpression of sFlt-1 as well as the addition of exogenous sFLT-1 (each binds and neutralizes VEGF) in mice attenuated lipopolysaccharide- and CLP-mediated mediated morbidity (cardiac dysfunction, vascular permeability and endothelial activation) and mortality in sepsis. Importantly, these findings have been reproduced and extended by others.6 The striking and reproducible reduction in morbidity and mortality make a compelling case for further exploration in human sepsis.

A role for Bevacizumab in treating patients with severe sepsis. There are several advantages in employing Bevacizumab as a lead agent for inhibiting VEGF signaling in patients with severe sepsis. First, as a humanized monoclonal antibody, it has a sufficiently long half-life that it may be given as a single injection in this patient population. Second, it is already FDA approved for use in patients with certain types of cancer. Thus, there is extensive knowledge of its pharmacokinetics and pharmacodynamics (at least in the latter population). Moreover, it should not be difficult to obtain permission for use in septic patients. Third, its chief side effect, namely hypertension, will not be a major concern in sepsis, since this condition is associated with hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are all adult patients, age > 18, who meet the following inclusion criteria:

  1. Evidence of infection a. temperature > 100.4F or < 97.0F of non-environmental causes, pneumonia as determined by the presence of an infiltrate on chest x-ray, a non-contaminated urinalysis with > 10 WBC or a urine dip-stick positive for leukocyte esterase, an abdominal CT scan yielding the diagnosis of an intra-abdominal etiology, skin/soft tissue infection on clinical exam.
  2. Two or more SIRS criteria a. tachycardia (HR>90) b. tachypnea (RR>20) or hypoxia (oxygen saturation<90%) c. hyperthermia >100.4 F (38C) or hypothermia <96F (35.5C) d. leukocytosis WBC> 15,000 cells/mm3 or bands>10%]
  3. Septic shock a. persistent hypotension (SBP < 90mmHg) after an initial 20-30 cc/kg fluid challenge, or the need for vasopressors for at least 1 hour in order to maintain a systolic blood pressure >90 mmHG; enrollment within 48 hours of meeting eligibility criteria.

Exclusion Criteria:

* Disease-Specific Exclusions:

  * Inability to obtain written informed consent from the patient or an appropriate designee General Medical Exclusions
  * Life expectancy of less than 12 weeks
* Bevacizumab-Specific Exclusions:

  * Inadequately controlled hypertension
  * Prior history of hypertensive crisis or hypertensive encephalopathy
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
  * History of myocardial infarction or unstable angina within 12 months prior to Day 1
  * History of stroke or transient ischemic attack within 12 months prior to Day 1
  * Known CNS malignancy, except for treated brain metastasis
  * Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
  * History of hemoptysis within 1 month prior to Day 1
  * History of chronic bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
  * Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
  * History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
  * Serious, non-healing wound, active ulcer, or untreated bone fracture
  * Proteinuria at screening
  * Known hypersensitivity to any component of bevacizumab
  * Pregnancy or lactation
  * Any clotting abnormalities or a history of deep venous thrombosis or pulmonary embolus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The change in Sequential Organ Failure Assessment score (SOFA) to assess reduction in organ failure | Between 0 and 72 hours

SECONDARY OUTCOMES:
Inflammation signaling: the change in circulating levels of IL-6 and TNF-alpha level as the primary | 1, 2, 3, 5, 7 and 28 days
Endothelial cell signaling/activation: change in E-selectin, ICAM-1, and sFLT | 1, 2, 3, 5, 7, 28 days
VEGF signaling: measurement of VEGF levels in response to the study drug or placebo and determine if there is a reduction in overall VEGF signaling. | 1, 2, 3, 5, 7, 28 days
Overall safety of Bevacizumab | Through Day 60
Mortality | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nathan I Shapiro, MD, Principal Investigator — Beth Israel Medical Center
Locations (3):
- United States (3):
  - Beth Israel Medical Center, Boston, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina

REFERENCES:
- [Derived] Shapiro NI, Aird WC. Sepsis and the broken endothelium. Crit Care. 2011 Mar 21;15(2):135. doi: 10.1186/cc10044. PMID 21457513